## **Consent form:**

| I | _have given my consent | for the participation i | n this research. | It is |
|---|---|---|---|---|
| investigating "the compariso | on between three differer | nt brushing techniques | for the reduction | n in |
| plaque accumulation" and | is being carried out b | у | The researcher | has |
| explained the purpose of t | the study and assured | me the confidentiality | y of the data. | The |
| researcher has given me the | right to withdraw from t | the study. | | |

## **Instructions:**

Participants will be instructed to refrain from brushing 2 days before their appointment to make sure proper plaque has been accumulated for removal. A trained dental student will carry out their brushing to ensure generalization.

## **Data collection instruments:**

Plaque index by Silness J and Loe H is being used in this study to assess the plaque removal by each tooth brushing technique.

The criterion for the index is:

| 0 | No plaque |
|---|---|
| 1 | A film of plaque adhering to the free gingiva margin and adjacent area of the |
| | tooth. The plaque may be recognized only after application of a disclosing |
| | agent or by running the explorer across the tooth surface. |
| 2 | Moderate accumulation of the soft deposits within the gingival pocket that |
| | can be seen with the naked eye or on the tooth and gingival margin. |
| 3 | Abundance of soft matter within the gingival pocket and/or the tooth and |
| | gingival margin. |

Patient name and signature:

**Doctors name and signature:**